CLINICAL TRIAL: NCT01500031
Title: Boston Scientific OffRoad™ Re-entry Catheter System for Subintimal Recanalization of Chronic Total Occlusions in Femoropopliteal Arteries
Acronym: Re-ROUTE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2273
Record Dates: First submitted 2011-12-19; First posted 2011-12-26 (Estimated); Results first posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Total Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OffRoad Re-entry catheter (Experimental): Participants treated with OffRoad Re-entry Catheter System
  Interventions: Device: OffRoad Re-entry Catheter System

INTERVENTIONS:
Device: OffRoad Re-entry Catheter System — Facilitate the placement and positioning of guidewires within the peripheral vasculature.

SUMMARY:
Study of the OffRoad™ Re-entry Catheter System for subintimal recanalization of chronic total occlusions in native femoropopliteal arteries.

ELIGIBILITY:
Inclusion Criteria:

* Claudication or critical limb ischemia (Rutherford Category 2-5)
* Documented de novo or re-occluded Chronic Total Occlusion (CTO) (99-100% stenosed) lesion in native femoropopliteal artery
* Target vessel occlusion length is ≥ 1 cm and ≤ 30 cm
* Minimum reference vessel diameter is 4 mm

Exclusion Criteria:

* Contraindication to an endovascular procedure
* Previous stent placement in the target vessel
* Prior surgery of the superficial femoral artery (SFA) in the target limb to treat atherosclerotic disease
* Platelet count <150,000 mm3 or >600,000 mm3
* Renal insufficiency with a serum creatinine >2.3 mg/dl
* History of major amputation (ankle level or above) in the same limb as the target lesion
* Current participation in another drug or device clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Schmidt, Principal Investigator — Herzzentrum Leipzig GmbH/ Park Krankenhaus Leipzig GmbH

REFERENCES:
- [Derived] Schmidt A, Keirse K, Blessing E, Langhoff R, Diaz-Cartelle J; European Study Group. Offroad re-entry catheter system for subintimal recanalization of chronic total occlusions in femoropopliteal arteries: primary safety and effectiveness results of the re-route trial. J Cardiovasc Surg (Torino). 2014 Aug;55(4):551-8. Epub 2014 Jun 13. PMID 24926886

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 92 subjects enrolled at 12 investigative centers in Belgium, Germany and Switzerland from 26 April 2012 to 16 April 2013
Groups:
- Re-ROUTE: All subjects who meet the inclusion criteria and are enrolled in this trial will be treated with the OffRoad™ Re-entry Catheter
Period: Overall Study
Arm/Group | Re-ROUTE
Started | 92
Completed | 87
Not Completed | 5
Not completed — Death | 1
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Re-ROUTE
Number analyzed (Participants) | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.29 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1
  Caucasian | 91
Region of Enrollment [Number; unit: participants]
  Belgium | 36
  Germany | 53
  Switzerland | 3
General Medical History [Number; unit: participants] — The same participant may be included in more than one category or not all participants may contribute to a category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    History of Smoking | 71
    Current Diabetes Mellitus | 47
    History of Hyperlipidemia requiring medication | 61
    History of Hypertension requiring medication | 75
    History of chronic obstructive pulmonary disease | 9
Cardiac History [Number; unit: participants] — The same participant may be included in more than one category or not all participants may contribute to a category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    History of Coronary Artery Disease | 30
    History of Myocardial Infarction | 16
    History of Congestive Heart Failure | 6
    Stable Angina | 2
    Unstable Angina | 0
    History of Percutaneous Coronary Intervention | 16
    History of Coronary Artery Bypass Graft | 5
Neurologic/Renal History [Number; unit: participants] — The same participant may be included in more than one category or not all participants may contribute to a category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    History of Transient Ischemic Attacks | 0
    History of Cerebrovascular Accident | 11
    History of Renal Insufficiency | 18
    History of Renal Percutaneous Intervention | 0
Peripheral Vascular History [Number; unit: participants] — The same participant may be included in more than one category or not all participants may contribute to a category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    History of Other Peripheral Interventions | 40
    History of Claudication | 82
Baseline Lesion Characteristics: Treated Limb [Number; unit: lesions]
  Right leg | 48
  Left leg | 44
Baseline Lesion Characteristics: Reference Vessel Diameter [Mean (Standard Deviation); unit: millimeters] | 5.18 (0.62)
Baseline Lesion Characteristics: % Occluded [Mean (Standard Deviation); unit: percentage Occluded] | 100.00 (0.00)
Baseline Lesion Characteristics: Lesion Length [Mean (Standard Deviation); unit: millimeters] | 175.12 (85.42)
Baseline Lesion Characteristics: Presence of Calcification [Number; unit: lesions] — Readily apparent densities seen within the artery wall and site of lesion as an x-ray-absorbing mass. The protocol does not provide the criteria for assessing lesions as "None/Mild", "Moderate", or "Severe". The assessment was left to the discretion of the Investigator.
  lesions
    None/Mild | 43
    Moderate | 44
    Severe | 5
Baseline Lesion Characteristics: Percent of Lesions with Re-entry into true lumen (site reported) [Number; unit: percent of lesions] — Re-entry in the true lumen defined as placement of a guidewire in the true lumen distal to a Chronic Total Occlusion (CTO).
  percent of lesions | 84.8
Baseline Lesion Characteristics: Percent of Lesions with Perforation requiring intervention [Number; unit: percent of lesions] — Perforation defined as Angiographic Perforation (Perforation detected by the clinical center or Angiographic Core Laboratory at any point during the procedure) or clinical Perforation (perforation requiring additional treatment (including efforts to seal the perforation), or resulting in significant hemodynamic compromise, abrupt closure, or death).
  percent of lesions | 4.3
Baseline Lesion Characteristics: Percent of Lesions with Flow limiting dissection [Number; unit: percent of lesions] — Type A: Small radiolucent area within vessel lumen disappearing with passage of contrast material, Type B: Appearance of contrast medium parallel to vessel lumen disappearing within a few cardiac cycles, Type C: Dissection protruding outside vessel lumen persisting after passage of contrast material, Type D: Spiral shaped filling defect with or without delayed run-off of contrast material in the antegrade flow, Type E: Persistent luminal filling defect with delayed run-off of contrast material in the distal lumen, Type F: Filling defect accompanied by total vessel occlusion.
  percent of lesions | 2.2
Procedural Characteristics: Primary diagnosis [Number; unit: participants]
  Claudication | 78
  Critical limb ischemia | 14
Procedural Characteristics: Urgency of intervention [Number; unit: participants]
  Emergent | 1
  Urgent | 3
  Elective | 88
Procedural Characteristics: Time from artery access to sheath removal [Mean (Standard Deviation); unit: minutes] | 87.51 (135.33)
Procedural Characteristics: Puncture site [Number; unit: participants]
  Right femoral | 49
  Right brachial | 0
  Left femoral | 42
  Left brachial | 0
  Other | 1
Procedural Characteristics: Total amount of contrast used [Mean (Standard Deviation); unit: milliliters] | 143.11 (74.57)
Procedural Characteristics: Total fluoroscopy time [Mean (Standard Deviation); unit: minutes] | 20.99 (13.10)
Procedural Characteristics: Number of participants with additional Vascular procedures performed [Number; unit: participants] | 50
Procedural Characteristics: Number of Participants with stent placement performed [Number; unit: participants] | 81
Procedural Characteristics: Number of Participants with other Devices used [Number; unit: participants] | 92
Procedural Characteristics: Number of non-target lesion treated [Mean (Standard Deviation); unit: lesions] — Additional non-target superficial femoral artery (SFA) lesions: e.g. carotid, renal, subclavian, iliac, opposite limb.
  lesions | 0.24 (0.52)
Procedural Characteristics: Number of Participants currently taking medication [Number; unit: participants] | 84

OUTCOME MEASURES:

1. Primary Outcome: Composite Rate of Major Adverse Events
Description: Composite rate of major adverse events (MAEs) related to the OffRoad System at 30 days, including: death, perforation requiring intervention, clinically significant peripheral embolism, and major amputation (amputation of the treated lower limb at the ankle level or above).
  Events are based on data adjudicated by a Clinical Event Committee.
Time Frame: 30 days
Population: The primary endpoints were analyzed on an intent-to-treat (ITT) basis. All subjects who signed and dated the written Informed Consent Form (ICF) and had any part of the OffRoad System introduced into the body were included in the ITT analysis. 2 participants were not evaluable (No follow-up ≥ 23 days and events-free within 30-day)
Measure: Number; unit: percentage of participants
Arm/Group | OffRoad Re-entry Catheter
Number analyzed (Participants) | 90
percentage of participants | 3.3

2. Primary Outcome: Effectiveness (On the Day of Procedure)
Description: Device Technical Success rate, defined as placement of a guidewire in the true lumen distal to a Chronic Total Occlusion (CTO)
Time Frame: Device technical success is determined during the index procedure, from the time of first puncture of the skin in order to obtain access to the artery until the time the introducer sheath is removed from the body
Population: The primary endpoints were analyzed on an intent-to-treat (ITT) basis. All subjects who signed and dated the written Informed Consent Form (ICF) and had any part of the OffRoad System introduced into the body were included in the ITT analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OffRoad Re-entry Catheter
Number analyzed (Participants) | 92
percentage of participants | 84.8 [77.4 to 92.1]

3. Other Pre Specified Outcome: Device-related Death
Description: All death related to the use of the OffRoad Re-entry Catheter System. Events are based on site reported Adverse Event data.
Time Frame: 30 days
Population: All subjects who signed and dated the written Informed Consent Form and had any part of the OffRoad System introduced into the body were included in the analysis. 2 participants were not evaluable (No follow-up ≥ 23 days and events-free within 30-day).
Measure: Number; unit: percentage of participants
Arm/Group | OffRoad Re-entry Catheter
Number analyzed (Participants) | 90
percentage of participants | 0.0

4. Other Pre Specified Outcome: Device-related Perforation Requiring Intervention
Description: All perforation requiring intervention related to the use of the OffRoad Re-entry Catheter System.
  Events are based on site reported Adverse Event data.
Time Frame: 30 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | OffRoad Re-entry Catheter
Number analyzed (Participants) | 90
percentage of participants | 0.0

5. Other Pre Specified Outcome: Device-related Clinically Significant Peripheral Embolism
Description: All clinically significant peripheral embolisms related to the use of the OffRoad Re-entry Catheter System.
  Events are based on site reported Adverse Event data.
Time Frame: 30 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | OffRoad Re-entry Catheter
Number analyzed (Participants) | 90
percentage of participants | 0.0

6. Other Pre Specified Outcome: Device-related Major Amputation at Ankle Level or Above of Treated Lower Limb
Description: All Major amputations related to the use of the OffRoad Re-entry Catheter System.
  Events are based on site reported Adverse Event data.
Time Frame: 30 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | OffRoad Re-entry Catheter
Number analyzed (Participants) | 90
percentage of participants | 0.0

7. Other Pre Specified Outcome: All Adverse Events
Description: All adverse events (AEs) reported by the centers.
Time Frame: 30 days
Population: as for outcome 3
Measure: Number; unit: adverse events
Arm/Group | OffRoad Re-entry Catheter
Number analyzed (Participants) | 90
adverse events | 46

8. Other Pre Specified Outcome: Acute Procedure Success
Description: Acute Procedure Success, defined as device technical success and the absence of in-hospital Major Adverse Events {death, perforation requiring intervention, clinically significant peripheral embolism, and major amputation (amputation of the treated lower limb at the ankle level or above)}
Time Frame: 30 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | OffRoad Re-entry Catheter
Number analyzed (Participants) | 90
percentage of participants | 73.3

9. Other Pre Specified Outcome: Target Lesion Revascularization Due to a Complication
Description: Any surgical or percutaneous intervention to the target lesion(s) after the index procedure.
Time Frame: 30 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | OffRoad Re-entry Catheter
Number analyzed (Participants) | 90
percentage of participants | 0.0

10. Other Pre Specified Outcome: Device-related Dissection, Grade C or Greater
Description: Type A- Small radiolucent area within the lumen of the vessel disappearing with the passage of the contrast material.
  Type B- Appearance of contrast medium parallel to the lumen of the vessel disappearing within a few cardiac cycles.
  Type C- Dissection protruding outside the lumen of the vessel persisting after passage of the contrast material.
  Type D- Spiral shaped filling defect with or without delayed run-off of the contrast material in the antegrade flow.
  Type E- Persistent luminal filling defect with delayed run-off of the contrast material in the distal lumen.
Time Frame: 30 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | OffRoad Re-entry Catheter
Number analyzed (Participants) | 90
percentage of participants | 0.0

11. Other Pre Specified Outcome: Overall Procedure Time
Description: Defined as the time when the treating physician first punctures the skin in order to obtain access to the artery to treat the target lesion until the time the introducer sheath is removed from the body.
Time Frame: On the day of Procedure
Population: All subjects who signed and dated the written Informed Consent Form and had any part of the OffRoad System introduced into the body were included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | OffRoad Re-entry Catheter
Number analyzed (Participants) | 92
minutes | 87.51 (135.33)

12. Other Pre Specified Outcome: OffRoad System Use Length of Time
Description: From time of "positioning balloon catheter" introduced in the body until time "final OffRoad component" removed.
Time Frame: On the day of Procedure
Population: All subjects who signed and dated the written Informed Consent Form and had any part of the OffRoad System introduced into the body were included in the analysis. 1 participant was not evaluable (No data available).
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | OffRoad Re-entry Catheter
Number analyzed (Participants) | 91
minutes | 11.14 (10.49)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | OffRoad Re-entry Catheter
Serious Adverse Events (participants affected / at risk) | 21/92
Other Adverse Events (participants affected / at risk) | 15/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OffRoad Re-entry Catheter (N=92)
Femoral artery dissection (Vascular disorders) | 2 (2)
Peripheral embolism (Vascular disorders) | 4 (4)
Femoral artery occlusion (Vascular disorders) | 2 (3)
Femoral arterial stenosis (Vascular disorders) | 2 (2)
Peripheral artery dissection (Vascular disorders) | 1 (1)
Arterial stenosis limb (Vascular disorders) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 1 (1)
Necrosis (General disorders) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Vascular injury (Injury, poisoning and procedural complications) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Preferred Term not coded (General disorders) | 1 (1) — System Class not coded
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OffRoad Re-entry Catheter (N=92)
Femoral artery dissection (Vascular disorders) | 4 (4)
Peripheral artery dissection (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Reperfusion injury (Vascular disorders) | 1 (1)
Oedema peripheral (General disorders) | 2 (2)
Catheter site haemorrhage (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator shall have the right to publish the results, provided that before publishing, the PI shall submit copies of any proposed publication or presentation to Sponsor for review at least 45 days in advance of submission for publication or presentation to a publisher or other third party. Sponsor reserves the right to delete any confidential information or other proprietary information of Sponsor from the proposed publication or presentation.